CLINICAL TRIAL: NCT05236127
Title: The Effect of Intermittent Fasting on Acute Subconcussive Head Impacts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Keisuke Kawata, Assistant Professor Kinesiology, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 13076
Record Dates: First submitted 2021-11-16; First posted 2022-02-11 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Sports Injury; Intermittent Fasting
Keywords: Soccer Heading; Subconcussive Head Impacts; Intermittent Fasting
MeSH Terms: conditions — Athletic Injuries; Intermittent Fasting

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The primary investigator will be blinded to the study participants' study group status. Additionally, the statistician will be blinded from group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Fasted (Experimental): Fasted Group: Individuals randomly assigned to undergo a 20 hour fast with a four hour eating window for the entire 8-day period of the study.
  Interventions: Other: Intermittent Fasting
- Pre-heading fasted (Experimental): Pre-Heading Fasted Group: Individuals randomly assigned to undergo a 20 hour fast with a 4 hour eating window for a 5-day period prior to the soccer heading.
  Interventions: Other: Intermittent Fasting
- Post-heading fasted (Experimental): Post-Heading Fasted Group: Individuals randomly assigned to undergo a 20 hour fast with a four hour eating window for a 3-day period following the soccer heading.
  Interventions: Other: Intermittent Fasting
- Control (Experimental): Control Group: Individuals randomly assigned to eat per usual over the course of the entire 8-day study period.
  Interventions: Other: Intermittent Fasting
- Subconcussive Head Impact (Active Comparator): All four groups undergo the same soccer heading model as described below.
  Device: Soccer Heading Soccer Heading: Subjects stood approximately 40 feet away from a JUGS soccer ball launcher and participated in 20 consecutive soccer headings, separated by 30 second intervals.
  Interventions: Other: Soccer Heading

INTERVENTIONS:
Other: Soccer Heading — A standardized and reliable soccer heading protocol will be used for the experiment. A triaxial accelerometer embedded in a head-band pocket and positioned directly below the external occipital protuberance (inion) to monitor linear and rotational head accelerations. A JUGS soccer machine will be used to simulate a soccer throw-in with a standardized ball speed of 25mph. The ball speed is similar to when soccer players make a long throw-in from the sideline to mid-field. Soccer players frequently perform this maneuver during practice and games. Subjects will stand approximately 40ft away from the machine to perform the heading. Participants perform 20 standing headers with 1 header per 30 seconds. The subjects will be instructed to direct the ball back toward the JUGS soccer machine in the air.
  Arms: Subconcussive Head Impact
Other: Intermittent Fasting — The purpose of this study is to examine the effect of intermittent fasting on the acute neural responses to subconcussive head impacts. The study is designed to identify the effects of 20 controlled soccer headings in college-aged soccer players in one of four groups (fasted, pre-fasted, post-fasted, or control) through the use of neural-injury blood biomarkers, magnetic resonance spectroscopy, functional, and diffusion MRI, and ocular-motor function across 4 acute time points. Participants will be randomly designed to one of the four groups which consist of an 8 day fast, 5 day fast, 3 day fast, or the non-fasted control group.
  Arms: Control; Fasted; Post-heading fasted; Pre-heading fasted

SUMMARY:
The purpose of this study is to examine the effect of intermittent fasting on the acute neural responses to subconcussive head impacts. The study is designed to identify the effects of 20 controlled soccer headings in college-aged soccer players in one of four groups (fasted, pre-fasted, post-fasted, or control) through the use of neural-injury blood biomarkers, magnetic resonance spectroscopy, functional, and diffusion MRI, and ocular-motor function across 4 acute time points. The central hypothesis is that the neuronal structural, physiological, and functional impairments from the subconussive head impacts will be lessened by intermittent fasting either before or after the soccer headings. The neural-injury blood biomarkers neurofilament light (NfL), glial fibrillary acidic protein (GFAP), Ubiquitin C-Terminal Hydrolase L1 (UCH-L1), and Tau will be measured in serum, with the hypothesis that fasting prior to the 20 soccer headings will result in a decreased heightened response compared to the post-heading fasted group and the controls. It is also hypothesized that repetitive subconcussive head impacts will impair neurocognitive function, as measured by regional changes in fMRI activation during a working memory task in the fasted groups. Twenty headings will significantly alter fMRI activation in the fasted groups from baseline. This impairment will not be observed in the control group. White matter microstructure will be measured by diffusion imaging metrics, with the hypothesis that 20 soccer headings will significantly disrupt microstructure in the fasted groups compared to baseline, but not in the control group. The study will also assess neuro-opthalmologic function as measured by the King-Devick test (KDT) and oculomotor function as measured by near-point-of-convergence (NPC) in response to subconcussive head impacts. The hypothesis is that NPC performance will be significantly impaired for longer than 24 hours in all the groups, but this impairment will be greater in the control group, and that the learning curve and expected improvement of KDT will be significantly blunted in both groups, with a display worsening in the control group.

DETAILED DESCRIPTION:
The researchers will use a randomized controlled trial design and recruit participants on a first-come, first-serve basis for the study. The four groups are; 8 day fast, 5 day pre-heading fast, 3 day post-heading fast, and control.

The study consists of 4 data collection time points in an 8-day period. The four data collection sessions will last approximately 2 hours. This study design will enable the researchers to test outcome measures over subacute and acute phases.

* On day 0. the 1st test session takes place immediately prior to the 8-day period.
* On day 4, the 2nd test session takes place right before the soccer heading.
* Participants will perform the soccer headers.
* On day 5, the 3rd test session takes place 24 hours after the soccer heading.
* On day 7, the 4th test session takes place 72 hours after the soccer heading.

When written informed consent is obtained, the researchers will use a self-reported health questionnaire to obtain demographic information. The information includes age, sex, race/ethnicity, years of soccer playing and heading experience, number and age of previous concussions, sleep habits, menstrual cycle, and diet history as well as assessment of other neurological conditions to screen participants' eligibility. Participants who meet the inclusion criteria and are free of exclusionary factors will advance to the testing procedures.

Soccer Heading:

A standardized and reliable soccer heading protocol will be used for the experiment. A triaxial accelerometer and gyroscope (Triax Technologies) embedded in a head-band pocket and positioned back of the head to monitor linear and rotational head accelerations. A JUGS soccer machine will be used to simulate a soccer throw-in with a standardized ball speed of 25mph across both groups. The ball speed is similar to when soccer players make a long throw-in from the sideline to mid-field. Soccer players frequently perform this maneuver during practice and game. Participants will stand approximately 40ft away from the machine to perform soccer ball headings. An average linear head acceleration from a header sits around 20 g, while regular corner or goal kicks (~50mph) yield accelerations above 50 g. Participants in all groups will perform 20 headers with 1 header per 30 seconds.

Questionnaires:

The researchers will also (1) assess depression, anxiety, stress and panic symptoms using the PHQ-9, GAD-7, and the Daily Stress Inventory; (2) alcohol use disorder using AUDIT; (3) cannabis use disorder using CUDIT; (4) mood states using POMS; and (5) concussion symptoms using SCAT.

Biological Impedance Assessment:

Body weight measures will be taken at each visit using a Bioelectrical Impedance Assessment (BIA, Tanita Corporation of America, Arlington Heights, IL). This is a method for estimating body composition, in particular body fat, muscle mass, and total body water composition. BIA uses a weak electric current flow through the body and the voltage is measured to calculate impedance (resistance) of the body.

NPC and KDT:

During each test session, various assessments will be conducted on each participant. First, ocular assessments consisting of near point of convergence (NPC) and the King-Devick Test (KDT) will be used to assessed ocular-motor function and neuro-ophthalmologic function, respectively. The NPC measures the closest point to which one can maintain convergence while focusing on an object before double vision occurs. Assessment will be repeated twice, and mean NPC scores will be used for statistical analyses. After they have finished NPC, participants will complete the KDT. The KDT assesses neuro-ophthalmologic function due to it's design of saccadic eye movements coupled with multiple facets of brain functions such as attention, language, and concentration. It will be administrated on a hand- held tablet. Participants will be given one trial "demonstration" card to practice the task. Following the demonstration card, participants will tap through 3 test cards. Participants will be asked to read aloud, left to right and top to bottom, a series of numbers on the test cards as fast and as accurate as they can while refraining from using his/her fingers as a reading guide. The 3 test cards progress in difficulty (i.e. guideline disappearance, numbers become more dense). The KDT records the total time, in seconds, participants spent to complete the task (all 3 test cards). Accuracy will be recorded by a lab personnel member who will stand behind the participant and record any errors (incorrect number, missed number, etc.) made during the testing.

Blood Biomarkers:

Antecubital vein blood draws will be performed each test session to help determine serum biomarker concentrations. A trained phlebotomist will thoroughly clean the inner elbow surface with an alcohol swab and draw 7 ml of whole blood into sterile Vacutainer tubes with 21G butterfly needle. After the blood draw, the participant will use gauze to maintain direct pressure and a bandage will be provided. Plasma will be assessed by the 4-plex Simoa assay platform (Quanterix), which is a magnetic bead-based ELISA that allows detection of biomarkers in femtomolar concentrations.

MRI Techniques:

Once completing the MRI screening procedure, participants will undergo the following standardized MRI protocols.

Diffusion tensor imaging (DTI) is the most widely used technique to study the microstructural integrity of white matter in vivo. DTI provides simple markers, such as mean diffusivity (MD) and fractional anisotropy (FA), that have been used to reflect microstructural tissue change during aging, neurological disorders, and traumatic brain injury (i.e., concussion). However, despite their sensitivity, MD and FA represent cellular diffusivity estimated by basic statistical descriptions that do not directly correspond to biophysiological parameters of the neural cellular integrity. DTI assumes Gaussian diffusion within a single microstructural compartment and thus has proven non-specific to axonal structural damage. To address this limitation, neurite orientation dispersion and density imaging (NODDI) has been characterized to assess microstructural integrity of axons using a non-Gaussian model with multiple compartments. NODDI allows researchers to measure axonal density within white matter, orientation of axonal dispersion, and free water diffusion. The combined approach using NODDI and DTI will uncover greater depth of progressive axonal degeneration in response to repetitive subconcussive head impacts.

Magnetic Resonance Spectroscopy data will be collected using a single-voxel PRESS (Point RESolved Spectroscopy) sequence. The researchers primary region of interest (ROI) for MRS analysis is the dorsolateral prefrontal cortex (DLPFC). This region plays a vital role in regulating memory, attention, emotion/behavior, and autonomic motor function, and previous studies have shown altered neurometabolic levels in this region after concussive and subconcussive injuries. The MRS voxel with a dimension of 15x20x25mm3 will be positioned in the DLPFC using the T1-weighted image as a reference. There will also be a MRS scan collected gathering information on the whole brain to compare to the single voxel scan of the DLPFC.

N-Back Task: The n-back task will be used to assess verbal (letters) memory. For the verbal n-back tasks, while in the scanner, participants will be presented a series of letters, with letters being displayed on the screen one at a time. Participants will be instructed to answer whether the target letter is the same or different from the letter presented, if it the presented target is the same or different from the letter presented 1-back or 2-back letters prior. If the target letter is the same, participants will be instructed to press the index button of the controller in their left hand and if the letter is different, participants will be instructed to press the index button of the controller in their right hand. The n-back task has a total duration of about 7 minutes.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 years of age
* At least three years of soccer heading experience

Exclusion Criteria:

* Diabetes
* Any current intermittent fasting or in the last 3-6 months
* Any head or eye injury 12 months prior to the study
* Any neurological disorders (e.g., seizures, closed head injuries with prolonged loss of consciousness (> 15 minutes), history of stroke, spinal cord/surgery)
* History of vestibular, ocular, or vision dysfunction
* Any injury that would prohibit the performance of soccer headings
* A history of eating disorder
* Any brain implants or recent surgeries with metal implants that prohibit undergoing an MRI
* Currently taking any medications affecting appetite
* Pregnant
* HIV

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-23 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Change in brain-derived blood biomarkers from day 4 to day 5 and group differences | Blood samples will be collected at day 4 (prior to heading) and day 5 (24 hours post-heading).
  Blood samples will be collected and centrifuged at 1500 x g for ten minutes at 4 degree celsius. Serum samples will be aliquoted and stored at -80 degree celsius until analysis.
  Serum samples will be assayed for neurofilament-light (NfL) and glial fibrillary acidic protein (GFAP). All expression levels in pg/mL.
Change in brain-derived blood biomarkers from day 4 to day 7 and group differences | Blood samples will be collected at day 4 (prior to heading) and day 7 (72 hours post heading).
  Blood samples will be collected and centrifuged at 1500 x g for ten minutes at 4 degree celsius. Serum samples will be aliquoted and stored at -80 degree celsius until analysis.
  Serum samples will be assayed for neurofilament-light (NfL) and glial fibrillary acidic protein (GFAP). All expression levels in pg/mL.
Change in regional fMRI activation during the memory task from day 4 to day 5 and group differences | fMRI procedures will be performed on day 4 (prior to heading) and day 5 (24 hours post-heading)
  A standardized MRI protocol acquired on a Siemens TIM Trio scanner, equipped with a 64 channel phased array head radiofrequency coil will be used to collect fMRI images while a working memory task is administered.
  The task based fMRI protocol consists of N-back verbal working memory and a resting state task.
Change in regional fMRI activation during the memory task from day 4 to day 7 and group differences | fMRI procedures will be performed on day 4 (prior to heading) and day 7 (72 hours post-heading)
  A standardized MRI protocol acquired on a Siemens TIM Trio scanner, equipped with a 64 channel phased array head radiofrequency coil will be used to collect fMRI images while a working memory task is administered.
  The task based fMRI protocol consists of N-back verbal working memory and a resting state task.
Change in regional resting state functional connectivity from day 4 to day 5 and group differences | fMRI procedures will be performed day 4 (prior to heading) and day 5 (24 hours post-heading).
  A standardized MRI protocol acquired on a Siemens TIM Trio scanner, equipped with a 64 channel phased array head radiofrequency coil will be used to collect resting state functional connectivity.
Change in regional resting state functional connectivity from day 4 to day 7 and group differences | fMRI procedures will be performed day 4 (prior to heading) and day 7 (72 hours post-heading).
  A standardized MRI protocol acquired on a Siemens TIM Trio scanner, equipped with a 64 channel phased array head radiofrequency coil will be used to collect resting state functional connectivity.
Change in axonal microstructure from day 4 to day 5 and group differences | MRI procedures will be performed day 4 (prior to heading) and day 5 (24 hours post-heading).
  A standardized MRI protocol acquired on a Siemens TIM Trio scanner, equipped with a 64 channel phased array head radiofrequency coil will be used to assess changes in diffusion metrics.
  Whole-brain Diffusion tensor imaging (DTI) will be performed with a multi-slice single-shot spin echo echoplanar pulse sequence (echo time [TE] = 81 ms; repetition time [TR] = 9 s) using 64 diffusion-encoding directions, isotopically distributed over the surface of a sphere with electrostatic repulsion.
Change in axonal microstructure from day 4 to day 7 and group differences | MRI procedures will be performed day 4 (prior to heading) and day 7 (72 hours post-heading).
  A standardized MRI protocol acquired on a Siemens TIM Trio scanner, equipped with a 64 channel phased array head radiofrequency coil will be used to assess changes in diffusion metrics.
  Whole-brain Diffusion tensor imaging (DTI) will be performed with a multi-slice single-shot spin echo echoplanar pulse sequence (echo time [TE] = 81 ms; repetition time [TR] = 9 s) using 64 diffusion-encoding directions, isotopically distributed over the surface of a sphere with electrostatic repulsion.
Change in a panel of metabolites from day 4 to day 5 and group differences | MRI procedures will be performed day 4 (prior to heading) and day 5 (24 hours post-heading).
  A standardized MRI protocol acquired on a Siemens TIM Trio scanner, equipped with a 64 channel phased array head radiofrequency coil will be used to assess changes in neurometabolic metrics. The metabolic panel includes the following: N-Acetylaspartate (NAA), Glutamine/Glutamate (Glx), Myo-Inositol (mI), Choline (Cho), and Creatine (Cr).
Change in a panel of metabolites from day 4 to day 7 and group differences | MRI procedures will be performed day 4 (prior to heading) and day 7 (72 hours post-heading).
  A standardized MRI protocol acquired on a Siemens TIM Trio scanner, equipped with a 64 channel phased array head radiofrequency coil will be used to assess changes in neurometabolic metrics. The metabolic panel includes the following: N-Acetylaspartate (NAA), Glutamine/Glutamate (Glx), Myo-Inositol (mI), Choline (Cho), and Creatine (Cr).

SECONDARY OUTCOMES:
Change in near point of convergence from day 0 to day 4 and group differences | Near point of convergence will be assessed at day 0 and day 4 (prior to heading).
  Participants will undergo a brief test of near-point of convergence
Change in near point of convergence from day 4 to day 7 and group differences | Near point of convergence will be assessed at day 4 (prior to heading) and day 7 (72 hours post-heading).
  Participants will undergo a brief test of near-point of convergence
Change in King Devick performance from day 0 to day 4 and group differences | King Devick performance will be assessed at day 0 and day 4 (prior to heading)
  Participants will undergo the King-Devick Test--a brief assessment of saccadic eye movements, attention, and visual and language processing
Change in King Devick performance from day 4 to day 7 and group differences | King Devick performance will be assessed at day 4 (prior to heading) and day 7 (72 hours post-heading).
  Participants will undergo the King-Devick Test--a brief assessment of saccadic eye movements, attention, and visual and language processing
Change in brain-derived blood biomarkers from day 0 to day 4 and group differences | Blood samples will be collected at day 0 and day 4 (prior to heading).
  Blood samples will be collected and centrifuged at 1500 x g for ten minutes at 4 degree celsius. Serum samples will be aliquoted and stored at -80 degree celsius until analysis.
  Serum samples will be assayed for neurofilament-light (NfL) and glial fibrillary acidic protein (GFAP). All expression levels in pg/mL.
Change in brain-derived blood biomarkers from day day 0 to day 5 and group differences | Blood samples will be collected at day 0 and day 5 (24 hours post heading).
  Blood samples will be collected and centrifuged at 1500 x g for ten minutes at 4 degree celsius. Serum samples will be aliquoted and stored at -80 degree celsius until analysis.
  Serum samples will be assayed for neurofilament-light (NfL) and glial fibrillary acidic protein (GFAP). All expression levels in pg/mL.
Change in brain-derived blood biomarkers from day day 0 to day 7 and group differences | Blood samples will be collected at day 0 and day 7 (72 hours post heading).
  Blood samples will be collected and centrifuged at 1500 x g for ten minutes at 4 degree celsius. Serum samples will be aliquoted and stored at -80 degree celsius until analysis.
  Serum samples will be assayed for neurofilament-light (NfL) and glial fibrillary acidic protein (GFAP). All expression levels in pg/mL.

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University School of Public Health, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
All study data will be included in publications.

REFERENCES:
- [Background] Anton SD, Moehl K, Donahoo WT, Marosi K, Lee SA, Mainous AG 3rd, Leeuwenburgh C, Mattson MP. Flipping the Metabolic Switch: Understanding and Applying the Health Benefits of Fasting. Obesity (Silver Spring). 2018 Feb;26(2):254-268. doi: 10.1002/oby.22065. Epub 2017 Oct 31. PMID 29086496
- [Background] Kawata K, Steinfeldt JA, Huibregtse ME, Nowak MK, Macy JT, Kercher K, Rettke DJ, Shin A, Chen Z, Ejima K, Newman SD, Cheng H. Association Between Proteomic Blood Biomarkers and DTI/NODDI Metrics in Adolescent Football Players: A Pilot Study. Front Neurol. 2020 Nov 16;11:581781. doi: 10.3389/fneur.2020.581781. eCollection 2020. PMID 33304306
- [Background] Nowak MK, Bevilacqua ZW, Ejima K, Huibregtse ME, Chen Z, Mickleborough TD, Newman SD, Kawata K. Neuro-Ophthalmologic Response to Repetitive Subconcussive Head Impacts: A Randomized Clinical Trial. JAMA Ophthalmol. 2020 Apr 1;138(4):350-357. doi: 10.1001/jamaophthalmol.2019.6128. PMID 32053162
- [Background] Koerte IK, Lin AP, Muehlmann M, Merugumala S, Liao H, Starr T, Kaufmann D, Mayinger M, Steffinger D, Fisch B, Karch S, Heinen F, Ertl-Wagner B, Reiser M, Stern RA, Zafonte R, Shenton ME. Altered Neurochemistry in Former Professional Soccer Players without a History of Concussion. J Neurotrauma. 2015 Sep 1;32(17):1287-93. doi: 10.1089/neu.2014.3715. Epub 2015 May 14. PMID 25843317